CLINICAL TRIAL: NCT01555255
Title: Malaria Rapid Diagnostic Tests (RDTs) in Pregnancy: Detection of Placental Malaria
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: UNICEF (Other); United Nations Development Programme (Unknown); World Bank (Other); World Health Organization (Other)
Responsible Party: Principal Investigator, Principal Investigator, Foundation for Innovative New Diagnostics, Switzerland
Other Study IDs: RPC390
Record Dates: First submitted 2012-03-14; First posted 2012-03-15 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2012-10

CONDITIONS: Malaria; Placental Malaria; Malaria in Pregnancy
Keywords: malaria; pregnancy; placental malaria; malaria in pregnancy; birth weight; anemia
MeSH Terms: conditions — Malaria; Birth Weight; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Red cell pellets, dried whole blood on filter paper, and fixed blood and placental tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
This study seeks to determine whether screening pregnant women for malaria with malaria rapid diagnostic tests (RDTs) may detect placental infection and predict risk of poor birth outcomes due to malaria in areas of varied malaria transmission in Africa.

DETAILED DESCRIPTION:
Malaria prevention measures for pregnant women are critical and available, but the effectiveness of intermittent preventive treatment (IPTp) with sulfadoxine-pyrimethamine, a cornerstone in this prevention effort, is declining with increasing parasite resistance. New drugs for IPTp are being considered, but there are disadvantages to presumptive use of the few remaining efficacious antimalarials. An alternative approach may involve screening with diagnostic tests to better target efficacious antimalarial treatment to asymptomatic women with laboratory evidence of malaria infection. Light microscopy of peripheral maternal blood misses a large proportion of cases, and PCR is unavailable in routine health care settings. Preliminary evidence suggests that detection of parasite antigen in peripheral blood may provide an accurate indicator of clinically significant infections and predict pregnancy outcomes. Therefore, screening with RDTs may offer an accurate and practical way to identify pregnant women who will benefit from targeted therapy for placental malaria infection. Antigen detection thresholds vary widely among RDTs, and the distribution of target antigens in peripheral blood circulation is expected to differ; therefore, the potential value of RDTs in this population can best be established by evaluating the detection of placental parasitemia for highly-characterized RDTs, enabling results to be extrapolated to other products and programs. The study described here is proposed to address this question.

ELIGIBILITY:
Specific participant selection criteria include:

1. Presenting for care after quickening and before onset of labor (i.e. in the second or third trimester of pregnancy)
2. Age between 16 years and 44 years, inclusive
3. Willingness and ability to follow up with study visits and activities through the duration of pregnancy and at delivery
4. Absence of history of serious adverse reaction to sulfa drugs
5. Absence of history of serious adverse reaction to artemisinin-based drugs (depending on national policy on treatment of malaria in pregnancy)
6. Absence of HIV infection (both because guidelines for malaria prevention in pregnancy for HIV-infected women differ from those for HIV-negative women, and in order to avoid confounding of pregnancy outcomes by HIV-related complications or treatments in this early evaluation)
7. Absence of history of or current obstetrical complications (e.g. pre-eclampsia, eclampsia, hypertension during pregnancy, post-partum hemorrhage, evidence of multiple gestation)
8. Absence of chronic disease (e.g. diabetes mellitus, sickle cell disease)
9. Absence of evidence of severe acute disease requiring inpatient management or referral
10. Provision of written informed consent
11. Enrollment Hb ≥7 g/dL

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women presenting for routine antenatal care in the second and third trimesters of pregnancy, at antenatal clinics at ≥2 sites of varied malaria transmission intensity in Africa
Sampling Method: Non-Probability Sample
Enrollment: 1205 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
accuracy of diagnostic tests during gestation | 2nd trimester of pregnancy
  accuracy of malaria RDTs, blood smears and PCR performed on maternal peripheral blood to diagnose or predict placental malaria during gestation
accuracy of diagnostic tests during gestation | 3rd trimester of pregnancy
  accuracy of malaria RDTs, blood smears and PCR performed on maternal peripheral blood to diagnose or predict placental malaria during gestation

SECONDARY OUTCOMES:
association of placental malaria with infant birth weight | at birth
association of placental malaria with maternal hemoglobin | twice during gestation and at delivery
accuracy of diagnostic tests at delivery | at delivery
  accuracy of malaria RDTs, peripheral blood smears and PCR performed on maternal peripheral blood to diagnose placental malaria at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Heidi A Hopkins, MD, Principal Investigator — Foundation for Innovative New Diagnostics, Kampala, Uganda; Jean-Bosco Ouedraogo, MD, PhD, Principal Investigator — IRSS, Direction Regionale de l'Ouest, Bobo-Dioulasso, Burkina Faso; David Bell, MBBS, PhD, Study Director — Foundation for Innovative New Diagnostics, Geneva, Switzerland; Jane Cunningham, MD, Study Director — UNICEF/UNDP/World Bank/WHO Special Programme for Research and Training in Tropical Diseases (TDR), Geneva, Switzerland; Miriam Nakalembe, MBChB, Principal Investigator — Makerere University Faculty of Medicine, Kampala, Uganda
Locations (2):
- IRSS, Direction Régionale de l'Ouest, Bobo-Dioulasso, Burkina Faso
- Tororo District Hospital, Tororo, Tororo District, Uganda

REFERENCES:
- [Derived] Canier L, Khim N, Kim S, Sluydts V, Heng S, Dourng D, Eam R, Chy S, Khean C, Loch K, Ken M, Lim H, Siv S, Tho S, Masse-Navette P, Gryseels C, Uk S, Van Roey K, Grietens KP, Sokny M, Thavrin B, Chuor CM, Deubel V, Durnez L, Coosemans M, Menard D. An innovative tool for moving malaria PCR detection of parasite reservoir into the field. Malar J. 2013 Nov 9;12:405. doi: 10.1186/1475-2875-12-405. PMID 24206649